CLINICAL TRIAL: NCT03555435
Title: Pilot Study of Standalone and Peer Supported Online Problem Solving Program in Veterans With Untreated Mental Health Problems
Brief Title: Pilot Study of Peer-Supported Online Problem-Solving Program
Acronym: PS-OPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PPO 16-323; HX-002361-01 (Other Grant/Funding Number: VA Health Services R & D)
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Results first posted 2020-12-16 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Problem-solving; Well-being; Peer Support; Online Mental Health Program
Keywords: Problem-solving; Stigma reduction; Peer support; Online mental health program

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with three groups: 1) Use of online problem-solving program on one's own. 2) Use of online problem-solving program with peer support. 3) Wait control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- On Your Own (Experimental): Participants in this group will use the online program on their own for 6 weeks.
  Interventions: Other: Moving Forward On Your Own
- Peer Support (Experimental): Participants in this group will use the online program on their own for 6 weeks with the support of a peer coach. Peer coaching sessions will consist of 6 15-20 minute sessions one time per week. Sessions will be guided by a Moving Forward Peer Support Manual.
  Interventions: Behavioral: Moving Forward with Peer Support
- Wait (Placebo Comparator): Participants in this group will wait 6 weeks.
  Interventions: Behavioral: Wait

INTERVENTIONS:
Other: Moving Forward On Your Own — Participants in this group will use the online program on their own for 6 weeks.
  Arms: On Your Own
Behavioral: Moving Forward with Peer Support — Participants in this group will use the online program on their own for 6 weeks with the support of a peer coach. Peer coaching sessions will consist of 6 15-20 minute sessions one time per week. Sessions will be guided by a Moving Forward Peer Support Manual.
  Arms: Peer Support
Behavioral: Wait — Participants in this group will wait 6 weeks.
  Arms: Wait

SUMMARY:
Many Veterans with mental health care needs go without care due to stigma, practical problems with getting services, and a high value on self-sufficiency. VHA has developed online programs aimed at fostering MH that are easy to access and may be more acceptable than psychotherapy. The purpose of this study is to learn whether peer-supported use of an online problem-solving course is acceptable and helpful and whether the study data can be collected online. Results of this pilot study would inform a larger study of the impact on problem-solving and mental health of a non-stigmatizing, online program - with and without peer support. If effective, peer supported online programs would improve the quality of care to Veterans with unmet mental health needs.

DETAILED DESCRIPTION:
Approval will be obtained from VA primary care staff leaders at Palo Alto Division and VA Palo Alto Community Based Outpatient Clinics (CBOCs) to mail notes and a study information card to patients who do not have stop codes for mental health or integrated care in their EMR records for the past six months. The study information cards will describe the study, how to enroll, and will direct the Veteran to REDCap eligibility screening questions. When eligibility is confirmed, REDCap will automatically alert research assistant to enroll participant and randomize.

Primary Care Mental Health Integration staff at each clinic may also refer patients to the study by entering referral information directly into secure, encrypted REDCap files or by handing the patient a study information card.

Community veterans will be invited via social media marketing. Ads will link to a study web site. Study web site will link potential participants to REDCap eligibility screening questions. When eligibility is confirmed, REDCap will automatically alert research assistant to enroll participant and randomize.

Veterans who decide to be in the study will be assigned by chance to one of three groups: An On Your Own group, a Peer Support group, or a Wait group. Veterans assigned to take the Moving Forward course with peer support or on their own will complete the course online and practice the problem-solving skills they learned for six weeks. Finishing the Moving Forward course takes a total of about four hours. Veterans in the peer support group will speak with a Veteran who is experienced with the course on the phone for 15 to 20 minutes once a week during the study about using the ideas and exercises in the course to solve problems. Veterans assigned to the wait group will answer questions online about problem-solving skills and their well-being at the start and after six weeks). They will be able to take the course if they would like to after the six weeks have passed. Veterans in the On Your Own and Peer Support groups will answer questions online at the beginning, middle, and end of the study about problem-solving skills, their opinions about the course and about peer support (if they got it), and their well-being. This will take 10 to 15 minutes each time.

ELIGIBILITY:
Inclusion Criteria:

* A Veteran of one of the U.S. military services, including National Guard and Reserves.
* Positive screen (score of 1 or more) on the PHQ-2 or GAD-2.
* Access to a phone and to a desktop or laptop computer with internet access.
* Willingness to be randomized to one of three conditions.
* Willingness to work with a Peer Support Specialist.

Exclusion Criteria:

* An active suicide plan.
* Changes in psychoactive medications in the past month.
* MH treatment in the past 6 months, including treatment from a PC-MHI team member.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eve Bernstein Carlson, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset containing IPD reported in a publication will be created and shared. Datasets meeting VA standards for disclosure to the public will be made available within 1 year of publication. Prior to distribution, a local privacy officer will certify that all datasets contains no PHI. Final data sets will be maintained locally until enterprise-level resources become available for long-term storage and access.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Datasets will be made available within 1 year of publication.
Access Criteria: Guidance on request and distribution processes will be provided by ORD. Those requesting data will be asked to sign a Letter of Agreement.

REFERENCES:
- [Derived] Possemato K, Wu J, Greene C, MacQueen R, Blonigen D, Wade M, Owen J, Keane T, Brief D, Lindley S, Prins A, Mackintosh MA, Carlson E. Web-Based Problem-solving Training With and Without Peer Support in Veterans With Unmet Mental Health Needs: Pilot Study of Feasibility, User Acceptability, and Participant Engagement. J Med Internet Res. 2022 Jan 13;24(1):e29559. doi: 10.2196/29559. PMID 35023846
- See also: Social media marketing ad with link to join the study — https://studypages.com/s/are-you-are-a-veteran-facing-challenging-problems-upgrade-your-problem-solving-skills-with-an-online-course-made-for-veterans-405563/
- See also: Link to REDCap eligibility screening questions — https://is.gd/MovingForwardCourse

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | On Your Own | Peer Support | Wait
Started | 28 | 27 | 26
Completed | 11 | 8 | 18
Not Completed | 17 | 19 | 8
Not completed — Lost to Follow-up | 17 | 19 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | On Your Own | Peer Support | Wait | Total
Number analyzed (Participants) | 28 | 27 | 26 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 24 | 26 | 76
  >=65 years | 2 | 3 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (10.3) | 54 (11.0) | 56 (9.4) | 54 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 14 | 33
  Male | 18 | 18 | 12 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 2 | 8
  Not Hispanic or Latino | 25 | 24 | 24 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2 | 4
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 4 | 8
  White | 22 | 20 | 18 | 60
  More than one race | 4 | 2 | 2 | 8
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 27 | 26 | 81

OUTCOME MEASURES:

1. Primary Outcome: Problem-Solving Skills, Knowledge, and Abilities Test
Description: The Problem-Solving Skills, Knowledge, & Abilities Test is a brief, multiple-choice test that measures mastery of the basic concepts and skills that are included in the Moving Forward program. Scores on the test can range from 0 to 12 with higher scores indicating greater problem-solving skills, knowledge, and abilities.
Time Frame: change from baseline to study end (6 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | On Your Own | Peer Support | Wait
Number analyzed (Participants) | 11 | 8 | 18
score on a scale | -.55 (1.64) | .38 (2.26) | -.17 (1.65)

2. Primary Outcome: Problem-Solving Confidence
Description: The Problem-Solving Confidence Test assesses participant's confidence in his/her own problem solving abilities. Scores on this measure can range from 0 to 9 with higher scores indicating greater problem-solving confidence.
Time Frame: change from baseline to study end (6 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | On Your Own | Peer Support | Wait
Number analyzed (Participants) | 11 | 8 | 18
score on a scale | 1.91 (1.97) | 2.63 (2.72) | 0.56 (1.72)

3. Secondary Outcome: GAD-7 Change
Description: The GAD-7 assesses the severity of anxiety symptoms associated with generalized anxiety in terms of the proportion of days assessed in which the symptoms were present. Score range 0-21. Positive values for change from baseline to study end represent decreases in anxiety. Negative values for change from baseline to end represent increases in anxiety.
Time Frame: change from baseline to study end (6 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | On Your Own | Peer Support | Wait
Number analyzed (Participants) | 11 | 8 | 18
score on a scale | 3.00 (4.80) | -0.87 (5.67) | 1.06 (4.26)

4. Secondary Outcome: Posttraumatic Stress Symptoms Change
Description: Symptom change was measured by 7 items from the Screen for Posttraumatic Stress Symptoms (SPTSS) and 4 items from the Dissociative Symptoms Scale (DSS). Scores for all items could range from 0 to 47. Scores on change could range from -47 to 47. Positive values for change from baseline to study end represent reductions in PTSD symptoms.
Time Frame: change from baseline to study end (6 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | On Your Own | Peer Support | Wait
Number analyzed (Participants) | 11 | 8 | 18
score on a scale | 4.55 (7.01) | 3.50 (9.09) | 1.89 (5.82)

5. Secondary Outcome: WHO-5 Well-Being Index Change
Description: The World Health Organization Well-Being Index (WHO-5) is a widely-used 5-item measure assessing subjective psychological well-being. Its design for use around the world and translation into 30 languages are indicative of its usefulness as a measure for a diverse population. Score range 0-25. Positive changes from baseline to study end represent decreases in well-being. Negative values for change from baseline to end represent increases in well-being.
Time Frame: change from baseline to study end (6 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | On Your Own | Peer Support | Wait
Number analyzed (Participants) | 11 | 8 | 18
score on a scale | -5.09 (4.30) | -3.12 (7.08) | -5.89 (5.51)

6. Secondary Outcome: PHQ-9 Change
Description: The PHQ-9 assesses the severity of depression in terms of the proportion of days assessed in which the symptoms were present. Score range 0-27. Positive values for change from baseline to end represent reductions in depression. Negative values for change from baseline to end represent increases in depression.
Time Frame: change from baseline to study end (6 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | On Your Own | Peer Support | Wait
Number analyzed (Participants) | 11 | 8 | 18
score on a scale | 2.82 (4.69) | -0.75 (6.63) | 1.61 (2.83)

7. Secondary Outcome: Client Satisfaction Questionnaire
Description: The Client Satisfaction Questionnaire (CSQ) is a standardized, widely-used measure of customer satisfaction with health services and programs. Total scores on the 7-items we used range from 7 to 28. Higher scores represent greater satisfaction.
Time Frame: at study end (6 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | On Your Own | Peer Support | Wait
Number analyzed (Participants) | 11 | 8 | 18
score on a scale | 22.9 (3.09) | 19.6 (6.09) | 17.9 (5.03)

8. Other Pre Specified Outcome: Stigma Measure (EZ-EASI)
Description: The Endorsed and Anticipated Stigma Inventory (EASI) is a tool for assessing different dimensions of stigma-related beliefs about mental health among military and veteran populations. Findings based on a national sample of U.S. veterans deployed in support of Operation Enduring Freedom (OEF) in Afghanistan or Operation Iraqi Freedom (OIF) in Iraq suggest that the EASI is a psychometrically sound instrument. Specifically, results revealed evidence for the internal consistency reliability, content validity, convergent and discriminant validity, and discriminative validity of EASI scales. Total scores on 13 items used range from 0 to 39. Higher scores represent greater endorsement of stigma-related beliefs.
Time Frame: measured once at baseline
Population: Data from this measure were available for all participants because it was administered with baseline measures at the time of enrollment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | On Your Own | Peer Support | Wait
Number analyzed (Participants) | 28 | 27 | 18
score on a scale | 12.5 (7.46) | 14.5 (8.36) | 15.7 (7.40)

9. Other Pre Specified Outcome: Moving Forward Usage
Description: Usage was assessed by total number of days logging in to online course Moving Forward. This data was collected daily and automatically during study participation.
Time Frame: daily for 6 weeks
Population: Data from this measure were available for all participants because they were collected automatically via programming that collected and reported log ins to use the course. The course was mounted on a learning management platform and participants were given anonymized links to access the course.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | On Your Own | Peer Support
Number analyzed (Participants) | 28 | 27
days | 1.2 (1.23) | 3.0 (4.52)

ADVERSE EVENTS:
Description: This study of an educational program was conducted entirely online or by phone and included no medical intervention, measures, or monitoring. Groups were assigned to benign educational interventions. Adverse Events are not monitored.
Arm/Group | On Your Own | Peer Support | Wait
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This was a pilot study primarily aimed at studying feasibility and acceptability of online study enrollment and data collection that was not powered to allow definitive conclusions from analyses. Study end measures were available from only 47% of participants randomized at baseline, indicating that online data collection is insufficient to obtain complete measures after the baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT03555435/Prot_SAP_000.pdf